CLINICAL TRIAL: NCT07203846
Title: Modulation of Gut Microflora With Rifaximin to Reduce High Platelet Reactivity in Post-Acute Coronary Syndrome Patients on Ticagrelor (FLORA-ACS)
Brief Title: Modulation of Gut MicroFLORA With Rifaximin to Reduce High Platelet Reactivity in Post-ACS Patients on Ticagrelor
Acronym: FLORA-ACS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Collaborators: Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Principal Investigator, Jacek Kubica, Prof., Collegium Medicum w Bydgoszczy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLORA-ACS
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: ACS - Acute Coronary Syndrome; Ticagrelor; Microbiota; Platelet Aggregation; Myocardial Infarction (MI); Blood Platelets; Drug Effects; Platelet Aggregation Inhibitors; Drug Resistance; Platelet Function Tests; Dysbiosis; Anti-Bacterial Agents; Rifaximin
Keywords: high platelet reactivity; HPR; Multiplate aggregometry; multiple electrode aggregometry; MEA; microbiome; gut flora; eubiotic; 16S rRNA sequencing; P2Y12 inhibitor
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Dysbiosis | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- High platelet reactivity patients receiving rifaximin (Experimental): Participants identified as having high platelet reactivity treated with oral rifaximine
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — Participants receiving a 7-day course of oral rifaximin 400 mg every 12 hours
  Other Names: Xifaxan

SUMMARY:
The FLORA-ACS study aims to evaluate the relationship between dysbiosis and high platelet reactivity during treatment with ticagrelor in patients with a history of acute coronary syndromes and investigate the use of rifaximin to eliminate dysbiosis and thus provide effective antiplatelet treatment.

DETAILED DESCRIPTION:
A research hypothesis has been formulated indicating dysbiosis of the gut microbiota as a possible cause of high platelet reactivity (HPR) during treatment with an antiplatelet agent, ticagrelor, in post-acute coronary syndrome (ACS) patients. The use of rifaximin, an antibiotic exhibiting an eubiotic effect, may correct gut dysbiosis and help determine whether changes in the microbiota influence HPR.

The FLORA-ACS study will enroll 50 subjects with a history of ACS treated with ticagrelor (standard maintenance dose of 90 mg orally twice a day) and characterized by HPR. Participants will be enrolled in the study no sooner than 1 month and no later than 12 months following the ACS incident.

Platelet activity will be tested using the multiple electrode aggregometry method (Multiplate analyzer) with the HPR defined based on the consensus paper of the Working Group on On-Treatment Platelet Reactivity. Concurrently, fecal samples will be collected for microbiome profiling. The microbiota will be analyzed in terms of fecal bacterial richness and diversity using 16S ribosomal RNA sequencing.

Participants will receive a 7-day course of oral rifaximin (400 mg every 12 hours). Both platelet activity and microbiota testing will be conducted at baseline and post-treatment. Additional laboratory testing will include complete blood count and C-reactive protein. An analysis of major adverse cardiovascular events (MACE) occurrence within a 6-month follow-up period is planned.

ELIGIBILITY:
Inclusion criteria:

* Between 18 and 80 years of age
* History of acute coronary syndrome no sooner than 1 month and no later than 12 months prior to study inclusion
* Current treatment with ticagrelor (90 mg orally twice a day)
* High platelet reactivity assessed with multiple electrode aggregometry method (AUC of >46 U)
* Provision of informed consent prior to any study procedures

Exclusion criteria:

* History of hypersensitivity to rifaximin or other rifamycin-derived agent
* Ongoing treatment with rifamycins
* Platelet count < 100×10^9/L or > 450×10^9/L
* Treatment with antibiotics, probiotics, or glucocorticoids within 3 months prior to study inclusion
* History of gastrointestinal diseases such as inflammatory bowel disease, bowel obstruction, or gastrointestinal tumor
* Infection, including gastrointestinal infection, within a month prior to study inclusion
* History of Clostridium difficile infection
* Current use of specific medications (warfarin, glycoprotein IIb/IIIa inhibitors, immunosuppressants, bile acid sequestrants, antidiarrheal agents)
* Impaired liver function classified as Child-Pugh class B or C
* Hemodynamic instability
* Pregnancy or breastfeeding
* Patients considered by the investigator to be uncooperative

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in platelet reactivity in Multiplate | 0-7 days
  Relative reduction in platelet reactivity from baseline to post-intervention by >10%, assessed with Multiplate analyzer (multiple electrode aggregometry)
Achievement of platelet reactivity below HPR | 0-7 days
  Achieving platelet reactivity below HPR in a patient with a higher baseline value, assessed with Multiplate analyzer (multiple electrode aggregometry)

SECONDARY OUTCOMES:
Relative reduction in platelet reactivity | 0-7 days
  Relative reduction in platelet reactivity from baseline to post-intervention by >10%, assessed with VerifyNow P2Y12 assay
Achieving platelet reactivity below HPR in VerifyNow | 0-7 days
  Achieving platelet reactivity below HPR in a patient with a higher baseline value, assessed with VerifyNow P2Y12 assay
Relative reduction in platelet reactivity in thromboelastography | 0-7 days
  Relative reduction in platelet reactivity from baseline to post-intervention by >10%, assessed with Platelet Mapping assay (thromboelastography)
Achieving platelet reactivity below HPR in thromboelastography | 0-7 days
  Achieving platelet reactivity below HPR in a patient with a higher baseline value, assessed with Platelet Mapping assay (thrombelastography)
Changes in microbiome profile | 0-7 days
  Changes in microbiome profile post-intervention assessed using 16S rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Kubica, Prof., Principal Investigator — Collegium Medicum w Bydgoszczy
Locations (1):
- Cardiology Department, Dr. A. Jurasz University Hospital, Bydgoszcz, Cuiavian-Pomeranian, Poland

IPD SHARING:
Plan to Share IPD: No